CLINICAL TRIAL: NCT01735253
Title: Metabolic Surgery for Type 2 Diabetes
Brief Title: Prospective Observatonal Study for Effect of Duodenojejunal Bypass and Gastric Bypass on T2DM Patients
Acronym: T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Inha University Hospital, IRB Inha University Hospital, Inha University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: inha 09-58
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Non Insulin Dependent Diabetes Mellitus
Keywords: metabolic surgery; gastric bypass; duodenojejunal bypass; type 2 DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gastric bypass, duodenojejunal bypass (Experimental)
  Interventions: Procedure: laparoscopic roux en Y gastric bypass / open duodenojejunal bypass

INTERVENTIONS:
Procedure: laparoscopic roux en Y gastric bypass / open duodenojejunal bypass — routine GBP with 80cm roux and biliopancreatic limb

SUMMARY:
Surgical treatment for type 2 diabetes has been taken note especially in less obese or non obese patients. In Asian, the nuber of less obses or non obese patients with T2DM is greater than that of the obese.

We are trying to do a prospective observational study for the evaluation of the effect of duidenojejunal bypass and gastric bypass on the glycemoc control in those patients.

The selection criteria are type 2 diabetess, 20-60 years old, BMI 23-34 or 21-22 with viceral obesity, insulin use less than 10 years and the patients understanding the hypothesis of this study, risks, expecting effects and agreeing this study.

We are checking oral GTT, insulin level, C-peptide level, HbA1C, etc. with some anthropometric measurs preoperatively, postoperatively, at 3 month and 12 month.

We will compare the clinical factors at each time.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* HbA1C > 7.0%
* BMI 23 - 34 or BMI 21-22 with viceral obesity
* insulin use less than 10 years
* uncerstanding the risks, hypothesis, expecting effects

Exclusion Criteria:

* type 1 diabetes
* C-peptide < 1.0ng/ml
* BMI < 21
* severe cardiovascular diseases or their history
* malignancy or history
* alcoholics, pituitary failrue
* history of severe ketosis, diabetic coma or precoma
* abnormal liver enzyme, over 3 fold of normal level
* liver cirrhosis or hepatitis
* serum creatinine > 2.0mg/dL
* glucocorticoids user
* diabetes due to other endocrine diseases
* pancreatic disease
* anti-GAD Ab (+)
* the incongruity for surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | preoperatively, at 3month, at 12 month
  change of the level

SECONDARY OUTCOMES:
oral glucose tolerance test | preopertively, postoperatively, at 3 month, at 12 month
  changes of the level at each time

OTHER OUTCOMES:
insulin level | preoperatively, postoperatively, at 3 month, at 12 month
  change the levels

CONTACTS AND LOCATIONS:
Locations (1):
- Yoonseok Heo, Incheon, South Korea